CLINICAL TRIAL: NCT04174833
Title: GlideScope Videolaryngoscopy in Patients With Reduced Mouth Opening, a Prospective Cohort Study
Brief Title: GlideScope Videolaryngoscopy in Patients With Reduced Mouth Opening
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Verathon (Industry)
Responsible Party: Sponsor
Other Study IDs: PV6094
Record Dates: First submitted 2019-10-06; First posted 2019-11-22 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Intubation;Difficult; Videolaryngoscopy; Small Mouth
Keywords: GlideScope; Airway Management; Videolaryngoscopic Intubation
MeSH Terms: conditions — Microstomia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to evaluate the clinical performance, quality of larynx visualization and difficulty of videolaryngoscopic intubation in patients with a reduced mouth opening (1.0 to 3.0 cm) utilizing the latest generation of GlideScopeTM Spectrum low profile laryngoscopy system.

DETAILED DESCRIPTION:
Reduced mouth opening in adults has been proven an important risk factor for difficult endotracheal intubation utilizing both direct and indirect laryngoscopy techniques, and a major reason for anesthesia-related adverse events. Over the past two decades, videolaryngoscopy has evolved to be the primary indirect laryngoscopy technique in a difficult endotracheal intubation setting. The possibility for optimal visualization of the laryngeal structures renders this method particularly helpful in patients with limited mouth opening. Especially videolaryngoscopy with acute-angle blades has been proposed to be favorable over conventional direct laryngoscopy in this setting. However, previous research has shown that a mouth opening of approximately 2.0 - 3.0 cm represents an independent risk factor and a possible critical lower limit for safe videolaryngoscopic intubation.

The latest generation of GlideScopeTM Spectrum blades may provide sufficient intubation conditions even in patients with a maximum mouth opening below 3.0 cm.

Our research group aims to evaluate the clinical performance, quality of larynx visualization and severity of videolaryngoscopic intubation the GlideScopeTM Spectrum system in patients with a small mouth opening.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for non-cardiac surgery
* Required general anesthesia and endotracheal intubation
* Mouth opening between 1.0 and 3.0 cm (any reason) recognized during preoperative assessment
* Written consent provided

Exclusion Criteria:

* Pregnant or breastfeeding women
* Confirmed indication for awake fiberoptic intubation, especially due to enoral and pharyngeal tumors, abscesses or other obstructive lesions
* Endotracheal intubation planned without deep general anesthesia or without neuromuscular blockade (e.g. awake videolaryngoscopy)
* Qualification for rapid sequence anesthesia induction due to risk of pulmonary aspiration
* Loose teeth

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients scheduled for non-cardiac surgery under general anesthesia with a need for endotracheal intubation presenting at the Anesthesiology Preassessment Clinic of the Hamburg University Hospital with a mouth opening between 1.0 and 3.0 cm within the recruiting period.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2021-11-17 (Actual)

PRIMARY OUTCOMES:
Successful videolaryngoscopic endotracheal intubation rate | Within 1 hour after anesthesia induction
  Observation during airway management

SECONDARY OUTCOMES:
First pass success rate | Within 1 hour after anesthesia induction
  Observation during airway management
Endotracheal intubation difficulty | Within 1 hour after concluded endotracheal intubation
  Subjective rating on a numeric rating scale [0-100]; 0 - very easy; 100 - very difficult
Best view obtained | Within 1 hour after concluded endotracheal intubation
  Cormack-Lehane classification
Intubation time | Within 1 hour after anesthesia induction
  Observation during airway management
Number of attempts | Within 1 hour after anesthesia induction
  Observation during airway management

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany